CLINICAL TRIAL: NCT02034825
Title: ASSESSing the Impact of Decipher on Practice Decision Making in Prostate Cancer After Surgery
Brief Title: Multi-site Decision Impact Study for Decipher
Acronym: ASSESS-D
Status: Completed | Type: Observational
Sponsor: GenomeDx Biosciences Corp (Industry)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: CU003
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2015-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Practicing urologic surgeons: * US board-certified
  * Practicing urologic surgeons
  * Performing at least 40 radical prostate surgeries annually
  Urologists will be excluded from participating in the study if:
  * They are unable to identify a the required number of eligible patient cases with available clinical data and tissue specimens;
  * They have spent less than 3 years in practice or perform less than 40 RP's per year
  All participants will be asked to complete a questionnaire based on a random selection of retroactively selected cases.
  Interventions: Other: Decipher Questionnaire

INTERVENTIONS:
Other: Decipher Questionnaire — Each participant will complete the pre and post-Decipher eCRQs for a minimum of 5 cases, and a maximum of 25 cases.

SUMMARY:
This prospectively designed retrospective clinical utility study will evaluate urologists' treatment recommendations before and after reviewing Decipher results for selected patient cases.

DETAILED DESCRIPTION:
The clinical utility of Decipher will be evaluated at two time-points:

1. Post RP - within 6 months after surgery
2. PSA rise - defined as PSA detectable and rising on 2 or more subsequent determinations

Patient cases will be retrospectively selected from at least 5 sites. Participating urologists at each site will be asked to each identify a minimum of 10 to a maximum of 50 suitable cases retrospectively. The resulting cases will then be de-identified, aggregated and evenly randomly distributed among the participating urologists via a secure on-line survey platform . All study participants (ie: urologists) will be masked to the original actual treatment decision and patient outcome.

The design of this study is such that any participating urologist may or may not review a patient originating from their own clinical practice, but will not review a case they themselves identified. Patient cases will be de-identified and randomized amongst participating urologists . By the retrospective nature of this study, cases may be several years post-RP. It is not expected that that participation in this study will have any impact on actual clinical management of patients.

Participants will be asked to complete two web-based electronic Case Report Questionnaires (eCRQ):

1. Pre-Decipher: will collect information on their recommended treatment decision and their decision confidence based on the de-identified clinical and pathological information provided for each patient case.
2. Post-Decipher: will collect their treatment recommendation and decision confidence for each de-identified patient case in the presence of the Decipher test results.

ELIGIBILITY:
Inclusion Criteria:

Patient cases eligible for this study were treated with radical prostatectomy and have one or more adverse features present as defined by AUA and NCCN guidelines:

* Pathological T3 stage of disease (i.e., ECE or SVI)
* Positive surgical margins, or
* Detectable PSA, defined as PSA detectable and rising on 2 or more subsequent determinations

Exclusion Criteria:

1. Metastatic Disease (M+) prior to surgery
2. Failure of PSA to nadir after surgery
3. Received any neo-adjuvant prostate cancer treatment before radical prostatectomy
4. Received any adjuvant chemotherapy
5. Required patient clinical data (Section 5.3) is not available for evaluation of eligibility criteria
6. Lack of documented treatment or management recommendation on file
7. Tissue specimen is inadequate for sampling and analysis

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient cases will be retrospectively selected from at least 5 sites. Participating urologists at each site will be asked to each identify a minimum of 10 to a maximum of 50 suitable cases retrospectively
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in treatment recommendation | 1.5 years
  Change in treatment recommendation from pre- to post-Decipher report, defined as any change in treatment recommendation. Specifically this will be defined as (pre- to post-):
  RT to ADT RT to ADT & RT RT to Observation ADT to RT ADT to ADT & RT ADT to Observation ADT & RT to RT ADT & RT to ADT ADT & RT to Observation Observation to RT Observation to ADT Observation to RT & ADT

SECONDARY OUTCOMES:
Specific change in treatment recommendation | 1.5 years
  1. Change in treatment recommendation from pre- to post-Decipher report defined as any of the following: Observation to Any treatment Any treatment to Observation
Changes in intensity of treatment | 1.5 years
  2. Change in treatment recommendation from pre- to post-Decipher report involving an increase or decrease in intensity defined as:
  • Increasing intensity: RT to ADT RT to ADT & RT ADT to ADT & RT Observation to any treatment
  • Decreasing intensity: Any treatment to observation ADT & RT to ADT ADT & RT to RT ADT to RT
Change in treatment recommendation compared to baseline | 1.5 years
  Changes in treatment recommendation (as described in the Primary Endpoint, and in Secondary Endpoints 1 and 2) from original, actual, treatment recommendation and post-Decipher recommendation.
Confidence in treatment recommendation | 1.5 years
  Changes in urologists expressed level of confidence in the treatment recommendation
Changes in the decision conflict scale | 1.5 years
Utility of Decipher | 1.5 years
  Urologist's perception regarding the utility of the Decipher test

CONTACTS AND LOCATIONS:
Overall Officials: Badani K Ketan, MD, Principal Investigator — Columbia University; Christine d Buerki, PhD, Study Director — GenomeDx Biosciences Inc.; Vipul Patel, MD, Principal Investigator — AdventHealth
Locations (3):
- United States (3):
  - Cedar Associates LLC, Menlo Park, California
  - Florida Hospital, Celebration, Florida
  - Columbia University, New York, New York

REFERENCES:
- [Background] Silberstein JL, Vickers AJ, Power NE, Fine SW, Scardino PT, Eastham JA, Laudone VP. Reverse stage shift at a tertiary care center: escalating risk in men undergoing radical prostatectomy. Cancer. 2011 Nov 1;117(21):4855-60. doi: 10.1002/cncr.26132. Epub 2011 Apr 11. PMID 21484780
- [Background] Thompson IM, Tangen CM, Paradelo J, Lucia MS, Miller G, Troyer D, Messing E, Forman J, Chin J, Swanson G, Canby-Hagino E, Crawford ED. Adjuvant radiotherapy for pathological T3N0M0 prostate cancer significantly reduces risk of metastases and improves survival: long-term followup of a randomized clinical trial. J Urol. 2009 Mar;181(3):956-62. doi: 10.1016/j.juro.2008.11.032. Epub 2009 Jan 23. PMID 19167731
- [Background] Bolla M, van Poppel H, Collette L, van Cangh P, Vekemans K, Da Pozzo L, de Reijke TM, Verbaeys A, Bosset JF, van Velthoven R, Marechal JM, Scalliet P, Haustermans K, Pierart M; European Organization for Research and Treatment of Cancer. Postoperative radiotherapy after radical prostatectomy: a randomised controlled trial (EORTC trial 22911). Lancet. 2005 Aug 13-19;366(9485):572-8. doi: 10.1016/S0140-6736(05)67101-2. PMID 16099293
- [Background] Wiegel T, Bottke D, Steiner U, Siegmann A, Golz R, Storkel S, Willich N, Semjonow A, Souchon R, Stockle M, Rube C, Weissbach L, Althaus P, Rebmann U, Kalble T, Feldmann HJ, Wirth M, Hinke A, Hinkelbein W, Miller K. Phase III postoperative adjuvant radiotherapy after radical prostatectomy compared with radical prostatectomy alone in pT3 prostate cancer with postoperative undetectable prostate-specific antigen: ARO 96-02/AUO AP 09/95. J Clin Oncol. 2009 Jun 20;27(18):2924-30. doi: 10.1200/JCO.2008.18.9563. Epub 2009 May 11. PMID 19433689
- [Background] Thompson IM Jr, Tangen CM, Paradelo J, Lucia MS, Miller G, Troyer D, Messing E, Forman J, Chin J, Swanson G, Canby-Hagino E, Crawford ED. Adjuvant radiotherapy for pathologically advanced prostate cancer: a randomized clinical trial. JAMA. 2006 Nov 15;296(19):2329-35. doi: 10.1001/jama.296.19.2329. PMID 17105795
- [Background] Schreiber D, Rineer J, Sura S, Teper E, Nabhani T, Han P, Schwartz D, Choi K, Rotman M. Radical prostatectomy for cT3-4 disease: an evaluation of the pathological outcomes and patterns of care for adjuvant radiation in a national cohort. BJU Int. 2011 Aug;108(3):360-5. doi: 10.1111/j.1464-410X.2010.09875.x. Epub 2010 Nov 18. PMID 21087395
- [Background] Badani K, Thompson DJ, Buerki C, Davicioni E, Garrison J, Ghadessi M, Mitra AP, Wood PJ, Hornberger J. Impact of a genomic classifier of metastatic risk on postoperative treatment recommendations for prostate cancer patients: a report from the DECIDE study group. Oncotarget. 2013 Apr;4(4):600-9. doi: 10.18632/oncotarget.918. PMID 23592338